CLINICAL TRIAL: NCT00433186
Title: Phase I, Open-label Study of Mycophenolate Mofetil In Systemic Sclerosis
Brief Title: Mycophenolate Mofetil in Systemic Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Aspreva Pharmaceuticals (Industry)
Responsible Party: Robert Lafyatis, MD, Boston University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-25973
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Mycophenolic Acid

ARMS (1):
- A (Experimental): Mycophenolate
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate 3000 mg each day
  Other Names: Cellcept

SUMMARY:
This is a research study of an investigational product called Mycophenolate mofetil (MMF). The study is designed to establish the safety and potential benefit of MMF. MMF has proven one of the most effective medications to date for SLE and associated nephritis. It also appears to be active in polymyositis and dermatomyositis. This medication inhibits inosine monophosphate dehydrogenase, the rate-limiting enzyme in synthesis of guanosine nucleotides. It blocks the type II isoform found in activated lymphocytes more potently than the type I isoform inhibiting both T- and B-lymphocytes. In SSc, MMF has been tried after anti-thymocyte globulin in one small open label study with efficacy with a significant improvement in skin score. We will test the safety and efficacy of MMF in SSc. All study patients will receive the study medication. The effect of the study medication will be examined in two subgroups of patients: those with early or progressive skin disease (skin substudy) and those with muscle disease (muscle substudy). The change in modified Rodnan skin score (MRSS) and creatinine phosphokinase (CK) for, respectively, the skin and muscle substudies at 6 months after treatment will be compared to baseline values.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is an autoimmune/connective tissue disease with complex pathogenesis involving immune system dysregulation, leading to fibrosis. Inflammatory and autoimmune aspects of this disease overlap systemic lupus erythematosus (SLE), a disease shown clearly to respond to MMF. Activated T-cells, the probable target of MMF in SLE, likely also play an important role in SSc pathogenesis. Evidence for this includes the similarity of SSc skin disease to chronic graft versus host disease, a disease in which T-cells play a critical role. MMF has proven one of the most effective medications to date for SLE and associated nephritis [1]. It also appears to be active in polymyositis and dermatomyositis, disease that also show significant overlap with SSc [2]. Myositis can also be a feature of SSc, suggesting that his disease manifestation might be particularly likely to respond to MMF. MMF inhibits inosine monophosphate dehydrogenase, the rate-limiting enzyme in synthesis of guanosine nucleotides. It blocks the type II isoform found in activated lymphocytes more potently than the type I isoform inhibiting both T- and B-lymphocytes [3]. In SSc, mycophenolate has been tried after anti-thymocyte globulin in one small open label study with efficacy with a significant improvement in skin score [4]. However, MMF has not been tried alone inSSc and has not been tried in muscle disease associated with SSc. In this study, we will test the safety and efficacy of MMF in SSc. In this study all study patients will receive the medication.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the American College of Rheumatology criteria for systemic sclerosis with diffuse cutaneous disease or muscle involvement
* Patients must also meet one of the following criteria:

SKIN SUBSTUDY (20 patients)

* Be within 1 1/2 years of first non-Raynaud's disease manifestation.
* How progression of skin disease at some time over the past 6 months prior to study entry based on either documented increase in skin score or new areas of skin involvement or progression (no more than 10 patients total recruited)

OR, MUSCLE SUBSTUDY (10 patients)

* Have a serum creatinine phosphokinase (CK) greater than 2 times the upper limit of normal

  * Patients entering the study on the basis of elevated CK must also have subjective and/or objective weakness; clinical evidence of cardiac, pulmonary or gastrointestinal disease as a complication of the patient¿s systemic sclerosis; or progressive skin disease.
  * The total number of patients entered in criteria 2a and 2b (skin substudy) will be 20. Patients meeting both criteria 2c. and either 2a or 2b will first be recruited into the muscle substudy (by criteria 2c) until 10 patients have been recruited.
  * Male or female patients >18 years of age.
  * Able and willing to give written informed consent and comply with the requirements of the study protocol
  * Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for 6 weeks after completion of treatment.
  * Adequate renal function as indicated by Cr less than or equal to 3.0
  * Adequate liver function, as indicated by SGOT and SGPT less than 2.5 times the upper limit of normal.
  * Negative serum pregnancy test (for women of child bearing age)

Exclusion Criteria:

* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer).
* Ongoing use of high dose steroids (>10mg/day) or unstable steroid dose in the past 4 weeks.
* Receipt of a live vaccine within 4 weeks prior to randomization.
* Previous Treatment with MMF
* Treatment with immunosuppressive, cytotoxic or anti-fibrotic drug within 4 weeks of screening other than anti-malarial. This includes cyclophosphamide, azathioprine (Immuran), methotrexate or other immunosuppressive or cytotoxic medication.
* Treatment with cholestyramine within 1 week of trial entry.
* History of HIV, Hepatitis B and/or Hepatitis C, or evidence of Hepatitis B or C at screening.
* Moderate to severe hepatic impairment, Child-Pugh Class B or C.
* History of recurrent significant infection or history of recurrent bacterial infections.
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* Active gastrointestinal bleeding within 4 weeks of study entry or active serious gastrointestinal disease.
* Pregnancy (a negative serum pregnancy test will be performed for all women of childbearing potential within 14 days of treatment).
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* A history of phenylketonuria, hereditary deficiency of hypoxanthine-guanine phosphoribosyl-transferase, Lesch-Nyhan or Kelley-Seegmiller syndrome
* Allergy to polysorbate 80/Tween
* Subjects who are breastfeeding
* Moderately severe renal dysfunction as indicated by Cr >3.0, dipstick protein >3+, or patient on dialysis.
* Hemoglobin: < 8.5 gm/dL
* Platelets: < 100,000/mm
* AST or ALT >2.5 x Upper limit of normal unless related to muscle disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Skin Study: The primary evaluation of response will be improvement of the modified Rodnan skin score @ 6 months. Improvement of skin score, correlates with improvement in joint function, functional status and physician's global assessment. | 6 months
Muscle Sub Study:The primary evaluation of response will be the CK at 6 months compared to baseline.Improvement after 6 months of tx compared to baseline CK will suggest efficacy | 6 months
Safety evaluation. | 6 months

SECONDARY OUTCOMES:
Secondary evaluations of response. Scleroderma Health Assessment Questionnaire (SHAQ): The SHAQ will be evaluated at study entry compared to 6 and 12 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lafyatis, MD, Principal Investigator — Boston University School od Medicine Rheumatology Section
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States